CLINICAL TRIAL: NCT04618120
Title: Comparison of Exercise Practices With Virtual Reality-based Exercise Training in Radiotherapy Period After Breast Cancer Surgery
Brief Title: Virtual Reality-based Exercise Training in Radiotherapy Period After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İlknur Onurlu, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2407471012
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Exercise; Upper Extremity Dysfunction
Keywords: Virtual Reality Exercises; Breast cancer; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality-based Exercise Group (Experimental): Virtual reality-based exercises, breathing exercises and patient education on general considerations.
  Virtual reality-based exercises were done using the "Microsoft Xbox 360 Kinect" system. Among the 'Kinect Sports' games, especially tennis, table tennis, boxing and bowling games including upper extremity movements were selected. These games require all-directional and repetitive motion of the shoulder and elbow joint. Patients played the games using the operated / affected side arms. Between games, the patient was rested in a chair. In the meantime, deep breathing exercises were done.
  The patients participated in virtual reality-based exercises 3 days a week (15-18 sessions in total) during the radiotherapy treatment continued (5-6 weeks). Each exercise session was set to last 30-40 minutes in total.
  Interventions: Other: Virtual reality-based exercise
- Exercise Group (Experimental): Stretching exercises, range of motion exercises, posture exercises, breathing exercises and patient education on general considerations.
  11 different exercises consisting of shoulder range of motion in all directions, stretching exercises, posture exercises and breathing exercises were performed in the presence of a physiotherapist.The patients participated in this exercise program 3 days a week (15-18 sessions in total) during the radiotherapy treatment continued (5-6 weeks). One session of the exercises was completed in an average of 30-40 minutes. The same exercises were repeated in each session.
  Interventions: Other: Exercise
- Control Group (No Intervention): Only patient education on general considerations.

INTERVENTIONS:
Other: Virtual reality-based exercise — Virtual reality-based exercises with "Microsoft Xbox 360 Kinect" and breathing exercises.
  Patient education
  Arms: Virtual Reality-based Exercise Group
Other: Exercise — Shoulder range of motion, stretching, posture and breathing exercises. Patient education
  Arms: Exercise Group

SUMMARY:
The main purpose of this study is to compare two different exercise approaches during the radiotherapy period in patients who have undergone breast cancer surgery.

DETAILED DESCRIPTION:
Exercise therapies are effective methods in the treatment of complications after breast cancer surgery. The study aims to compare exercise practices with virtual reality-based exercise training during radiotherapy period after breast cancer surgery. Patients were randomly divided into 3 groups as virtual reality group, exercise group, and control group, considering the order of arrival at the clinic and the type of surgery (mastectomy and breast-conserving surgery). Patients in virtual reality group received virtual reality-based exercise training using Microsoft Xbox 360 Kinect (Redmond, WA). Patients in exercise group received an exercise program including range of motion, posture, stretching and breathing exercises. Both exercise groups participated in the exercise program for 30- 40 minutes, 3 days a week, as long as radiotherapy continued (5-6 weeks). Patients in the control group did not receive any exercise intervention as is done in the current practice. Assessment methods were applied at the beginning and at the end of the radiotherapy for all groups. Shoulder range of motion was measured using universal goniometer. Hand grip strength was measured using Jamar hand dynamometer. Shoulder proprioception was measured using Cybex (Lumex,NY,USA) isokinetic dynamometer. Upper extremity functional status, kinesiophobia, anxiety and depression level, fatigue and quality of life were evaluated with various questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being literate
* Having a diagnosis of unilateral breast cancer
* Having undergone surgery for breast cancer
* Radiotherapy will be applied for breast cancer treatment.

Exclusion Criteria:

* Metastasis
* Have an active infection
* Having a cardiac or neurological disease that would prevent participation in the study
* Having uncontrolled hypertension
* Having an orthopedic disorder that prevents exercise
* Having sensory or cognitive impairments that interfere with communication

Ages: 28 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Change in the shoulder range of motion | Baseline and after the exercise training (5-6 weeks)
  Universal Goniometer
Change in the grip strength assessed by hydraulic hand dynamometer | Baseline and after the exercise training (5-6 weeks)
  Jamar Hydraulic Hand Dynamometer
Change in the shoulder proprioception assessed by isokinetic dynamometer | Baseline and after the exercise training (5-6 weeks)
  Cybex 770 Norm isokinetic dynamometer (Lumex Inc. NY,USA)
Change in circumference of upper extremities | Baseline and after the exercise training (5-6 weeks)
  Lymphedema circumference measurement
Change in the functionality of upper extremities assessed by the Disability of Arm, Shoulder and Hand Questionnaire | Baseline and after the exercise training (5-6 weeks)
  The Turkish version of the Disability of Arm, Shoulder and Hand Questionnaire is used to evaluate functional status of upper extremities. The questionnaire consists of 30 questions. A score between 0-100 is obtained from the questionnaire. 0 point means "no disability", 100 point means "maximum level of disability".
Change in kinesiophobia assessed by theTampa Kinesiophobia Scale | Baseline and after the exercise training (5-6 weeks)
  The Turkish version of theTampa Kinesiophobia Scale was used to determine the level of kinesiophobia. 4-point Likert scoring (1 = Strongly disagree, 4 = Strongly agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. A score between 17-68 is obtained from the scale. The higher scores indicate higher kinesiophobia level.
Change in anxiety and depression level assessed by the Hospital Anxiety and Depression Scale | Baseline and after the exercise training (5-6 weeks)
  The Turkish version of the Hospital Anxiety and Depression Scale was used to determine the anxiety and depression level. The scale consists of 14 questions in total. 7 of the questions measure depression, 7 measure anxiety. A total score between 0-42 is obtained from the sum of the anxiety and depression scores. The higher scores indivate higher depression and /or anxiety.
Change in fatigue assessed by Piper Fatigue Scale | Baseline and after the exercise training (5-6 weeks)
  The Turkish version of Piper Fatigue Scale was used to determine the level of fatigue. The scale consists of 22 items (0-10 points) and 4 subscales: behavioral/severitiy (6 items), affective meaning (5 items), sensory (5 items) and cognitive/mood (6 items). Each subscale is scored individually and then aggregated together for an overall score. Higher scores indicate more fatigue.
  As a result of the average score; 0 points are interpreted as no fatigue, 1-3 points mild fatigue, 4-6 points moderate fatigue, 7-10 points severe fatigue.
  There are also 5 more questions in the scale that are not used in the subscale or total score calculation. These open-ended questions are about the duration of perceived fatigue, its causes, methods to alleviate fatigue and associated symptoms. They provide qualitative data.
Change in quality of life assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline and after the exercise training (5-6 weeks)
  The Turkish version of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) was used to evaluate quality of life level. It contains five functioning scales (physical, social, role, cognitive, and emotional functioning), eight symptom scales (fatigue, nausea/vomiting, pain, dyspnea, sleep disturbances, appetite loss, constipation, and diarrhea), financial impact, and overall quality of life. All scale scores are converted to range from 0 to 100. higher scores indicate better functioning for the functioning scales and overall quality of life; higher scores indicate higher symptom burden for the symptom scales.

SECONDARY OUTCOMES:
Patient Satisfaction | Patient satisfaction was evaluated at the end of the 5-6 week exercise training.
  The motivation of the exercises, the state of enjoying the exercise, believing that the exercise is beneficial, and the patient's willingness to continue the exercise were evaluated with 4 questions that they could answer with Likert-type answers.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Onurlu, PhD, Principal Investigator — Gazi University Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Emek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No